CLINICAL TRIAL: NCT06957808
Title: Investigating the Effect of Diroximel Fumarate on Glutathione in Schizophrenia
Acronym: FORTUNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Rosetrees Trust (Other)
Responsible Party: Principal Investigator, Katherine Beck, Dr, King's College London
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 331465
Record Dates: First submitted 2025-05-02; First posted 2025-05-05 (Actual); Last update posted 2025-05-05 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia Disorders
Keywords: psychosis; schizophrenia; inflammation; diroximel fumarate; neuroimaging; antioxidant; glutathione
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Inflammation | interventions — diroximel fumarate

STUDY DESIGN:
Intervention Model Description: Open label for 2 weeks then randomised to placebo or active drug for further 2 weeks
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Open label (Experimental): Participants take the research drug for 14 days in an open label phase.
  Interventions: Drug: Diroximel fumarate (DRF)
- Double-blind - DRF (Active Comparator): After open label phase, participants can be randomised to either the research drug (diroximel fumarate, DRF) or placebo for a further 2 weeks.
  Interventions: Drug: Diroximel fumarate (DRF)
- Double blind - Placebo (Placebo Comparator): After open label phase, participants can be randomised to either the research drug (diroximel fumarate, DRF) or placebo for a further 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diroximel fumarate (DRF) — Diroximel fumarate is an immunomodulating drug licensed for use in multiple sclerosis. It has been found to cross the blood brain barrier and increase brain glutathione levels.
  Other Names: Vumerity
  Arms: Double-blind - DRF; Open label
Drug: Placebo — A placebo pill given to participants.
  Arms: Double blind - Placebo

SUMMARY:
Schizophrenia is a condition that causes symptoms like delusions, hallucinations, reduced motivation and muddled thinking. It is a common, severe and disabling psychiatric illness affecting about 1/100 (1%) of people. It is ranked the third most disabling illness worldwide. Six in seven patients do not recover from the illness in 6-12 months and continue to experience psychotic symptoms. Therefore, there is a strong unmet need for new evidence-based treatments to target the neurobiology underlying schizophrenia. There is increasing evidence to indicate that glutathione (GSH), the main brain antioxidant, is abnormal in schizophrenia and may provide a new treatment target. In this study we plan to determine whether Diroximel Fumarate (DRF) (currently a treatment for a brain disorder called multiple sclerosis) can increase GSH in the brain of patients with schizophrenia using a brain scan (MRI) and explore whether changes in GSH are related to other brain measures (measured with MRI and EEG- which measures electrical activity in the brain), blood markers of GSH, and symptoms. During this study 30 people with schizophrenia will be recruited. They will take the drug DRF for two weeks, a computer will then decide randomly whether each person will continue to take DRF or a placebo/dummy pill for another two weeks. During this part of the study neither the patients nor the researchers will know which type of drug the patient is taking. Brain GSH and the other measures described will be assessed before and after taking the DRF and placebo/dummy pill. At the end of the study (2027), we will see if taking DRF alters the brain chemical (GSH) in people with schizophrenia and whether this is linked to other measures and symptoms. It will also give researchers information about the best way to design future studies for patients with schizophrenia using this drug.

DETAILED DESCRIPTION:
Study Objectives: To determine if the level of GSH in the ACC, as indexed by 1HMRS, will increase after treatment with DRF compared to baseline in patients with schizophrenia.

Study Design: Participants will take DRF as open label for 2 weeks (231mg for 7 days, then increase to 462mg for another 7 days), then they will have the option to participate in the second phase of the study, where they will be randomly allocated to either DRF for further 2 weeks or placebo. Allocation will be double-blinded. Participants will have baseline blood tests, schizophrenia rating scales, EEG and MRI, and these will be repeated after the open label and once again after the randomised phase.

30 patients with schizophrenia will be recruited from mental health teams.

Inclusion Criteria:

* 18-65 years
* diagnosis of schizophrenia (Diagnostic and Statistical Manual of Mental Disorders-5 (SCID) (DSM-5)
* stable antipsychotic dose (no change for 1 month)
* currently stable in mental state with no evidence of relapse within the last 2 months prior to study enrolment
* minimum score of 60 Positive and Negative Syndrome Scale (PANSS)
* capacity to provide informed consent

Exclusion criteria (https://www.medicines.org.uk/emc/product/13087/smpc):

* history of significant co-morbid medical or neurological disorder including but not limited to HIV, malignancies, Systemic Lupus Erythematosus, sarcoidosis, autoimmune vasculitis, bone marrow transplantation
* current use of medication that is known to interact with DRF, live vaccines given within the period of DRF treatment, nephrotoxic medication (including but not limited to aminoglycosides, diuretics, non-steroidal anti-inflammatory drugs, Lithium)
* contraindications to DRF (pregnancy, women of childbearing potential not currently using effective contraception (combined pill (oestrogen & progesterone), progesterone -only with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, sexual abstinence), breast feeding, severe hepatic impairment, moderate renal impairment, severe active gastrointestinal disease, lymphocyte count - below the Lower Limit of Normal (LLN) for the local laboratory (e.g 1.30 x109/L LLN for Viapath Kings College London), suspected or confirmed progressive multifocal leukoencephalopathy (PML), presence of risk factors for PML (previous and/or current immunosuppressant or immunomodulatory treatment (including natalizumab, other fumaric esters including Dimethyl Fumarate (DMF) (topical or systemic)), serious infection, current or recent herpes virus infection)
* substance dependence/abuse other than to cigarettes
* current high suicide risk
* participation in a clinical study of unlicensed medicines within the previous 30 days
* presence/history of other acute or chronic illness that would make participating unsafe or unsuitable, any contraindication to MRI scanning (e.g. claustrophobia, metallic implants, pacemaker, vascular clips, metal in eyes, pregnancy)
* allergies to any of DRFs ingredients
* taking part in a research study involving an unlicensed medicine within the last 30 days

ELIGIBILITY:
Inclusion Criteria:

* 18 -65 years, diagnosis of schizophrenia (Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
* Stable antipsychotic dose (no change for 1 month)
* Currently stable with no evidence of relapse within the last 2 months prior to study enrolment
* Minimum of 60 on the Positive and Negative Syndrome Scale (PANSS)
* Capacity to provide informed consent

Exclusion Criteria:

* History of significant co-morbid medical or neurological disorder including but not limited to HIV, malignancies, Systemic Lupus Erythematosus, sarcoidosis, autoimmune vasculitis, bone marrow transplantation
* Current use of medication that is known to interact with DRF, live vaccines given within the period of DRF treatment, nephrotoxic medication (including but not limited to aminoglycosides, diuretics, non-steroidal anti-inflammatory drugs, Lithium)
* Contraindications to DRF (pregnancy, women of childbearing potential not currently using effective contraception (combined pill (oestrogen & progesterone), progesterone -only with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, sexual abstinence), breast feeding, severe hepatic impairment, moderate renal impairment, severe active gastrointestinal disease, lymphocyte count - below the Lower Limit of Normal (LLN) for the local laboratory (e.g 1.30 x109/L LLN for Viapath King's College London), suspected or confirmed progressive multifocal leukoencephalopathy (PML), presence of risk factors for PML (previous and/or current immunosuppressant or immunomodulatory treatment (including natalizumab, other fumaric esters including Dimethyl Fumarate (DMF) (topical or systemic)), serious infection, current or recent herpes virus infection)
* Substance dependence/abuse other than to cigarettes
* Current high suicide risk
* Participation in a clinical study of unlicensed medicines within the previous 30 days
* Presence/history of other acute or chronic illness that would make participating unsafe or unsuitable, any contraindication to MRI scanning (e.g. claustrophobia, metallic implants, pacemaker, vascular clips, metal in eyes, pregnancy)
* Allergies to any of DRFs ingredients
* Taking part in a research study involving an unlicensed medicine within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
MRS glutathione (GSH) levels in ACC | Within one year of conclusion of the Research
  Glutathione levels in the Anterior Cingulate Cortex (ACC) measured by magnetic resonance spectroscopy (1HMRS)

SECONDARY OUTCOMES:
MMN Amplitude | Within one year of conclusion of the Research
  Mismatch negativity Amplitude measured by electroencephalography (EEG)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Beck, Clinical Lecturer, Principal Investigator — Department of Psychosis Studies, Institute of Psychiatry, Psychology and Neuroscience
Locations (3):
- United Kingdom (3):
  - South London and Maudsley NHS Foundation Trust, London, Greater London
  - Department of Computer Science, Faculty of Engineering Science, University College London, London, Greater London
  - School of Psychology, University of birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawryluk JW, Wang JF, Andreazza AC, Shao L, Young LT. Decreased levels of glutathione, the major brain antioxidant, in post-mortem prefrontal cortex from patients with psychiatric disorders. Int J Neuropsychopharmacol. 2011 Feb;14(1):123-30. doi: 10.1017/S1461145710000805. Epub 2010 Jul 16. PMID 20633320
- [Background] Ustun TB, Rehm J, Chatterji S, Saxena S, Trotter R, Room R, Bickenbach J. Multiple-informant ranking of the disabling effects of different health conditions in 14 countries. WHO/NIH Joint Project CAR Study Group. Lancet. 1999 Jul 10;354(9173):111-5. doi: 10.1016/s0140-6736(98)07507-2. PMID 10408486
- [Background] Raffa M, Mechri A, Othman LB, Fendri C, Gaha L, Kerkeni A. Decreased glutathione levels and antioxidant enzyme activities in untreated and treated schizophrenic patients. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Oct 1;33(7):1178-83. doi: 10.1016/j.pnpbp.2009.06.018. Epub 2009 Jul 2. PMID 19576938
- [Background] Owjfard M, Karimi F, Mallahzadeh A, Nabavizadeh SA, Namavar MR, Saadi MI, Hooshmandi E, Salehi MS, Zafarmand SS, Bayat M, Karimlou S, Borhani-Haghighi A. Mechanism of action and therapeutic potential of dimethyl fumarate in ischemic stroke. J Neurosci Res. 2023 Sep;101(9):1433-1446. doi: 10.1002/jnr.25202. Epub 2023 May 14. PMID 37183360
- [Background] Linker RA, Lee DH, Ryan S, van Dam AM, Conrad R, Bista P, Zeng W, Hronowsky X, Buko A, Chollate S, Ellrichmann G, Bruck W, Dawson K, Goelz S, Wiese S, Scannevin RH, Lukashev M, Gold R. Fumaric acid esters exert neuroprotective effects in neuroinflammation via activation of the Nrf2 antioxidant pathway. Brain. 2011 Mar;134(Pt 3):678-92. doi: 10.1093/brain/awq386. PMID 21354971
- [Background] Jauhar S, Veronese M, Nour MM, Rogdaki M, Hathway P, Turkheimer FE, Stone J, Egerton A, McGuire P, Kapur S, Howes OD. Determinants of treatment response in first-episode psychosis: an 18F-DOPA PET study. Mol Psychiatry. 2019 Oct;24(10):1502-1512. doi: 10.1038/s41380-018-0042-4. Epub 2018 Apr 20. PMID 29679071
- [Background] Jaaskelainen E, Juola P, Hirvonen N, McGrath JJ, Saha S, Isohanni M, Veijola J, Miettunen J. A systematic review and meta-analysis of recovery in schizophrenia. Schizophr Bull. 2013 Nov;39(6):1296-306. doi: 10.1093/schbul/sbs130. Epub 2012 Nov 20. PMID 23172003
- [Background] Halstead S, Siskind D, Amft M, Wagner E, Yakimov V, Shih-Jung Liu Z, Walder K, Warren N. Alteration patterns of peripheral concentrations of cytokines and associated inflammatory proteins in acute and chronic stages of schizophrenia: a systematic review and network meta-analysis. Lancet Psychiatry. 2023 Apr;10(4):260-271. doi: 10.1016/S2215-0366(23)00025-1. Epub 2023 Feb 27. PMID 36863384
- [Background] Gysin R, Kraftsik R, Sandell J, Bovet P, Chappuis C, Conus P, Deppen P, Preisig M, Ruiz V, Steullet P, Tosic M, Werge T, Cuenod M, Do KQ. Impaired glutathione synthesis in schizophrenia: convergent genetic and functional evidence. Proc Natl Acad Sci U S A. 2007 Oct 16;104(42):16621-6. doi: 10.1073/pnas.0706778104. Epub 2007 Oct 5. PMID 17921251
- [Background] Gold R, Arnold DL, Bar-Or A, Fox RJ, Kappos L, Mokliatchouk O, Jiang X, Lyons J, Kapadia S, Miller C. Long-term safety and efficacy of dimethyl fumarate for up to 13 years in patients with relapsing-remitting multiple sclerosis: Final ENDORSE study results. Mult Scler. 2022 Apr;28(5):801-816. doi: 10.1177/13524585211037909. Epub 2021 Sep 1. PMID 34465252
- [Background] Do KQ, Trabesinger AH, Kirsten-Kruger M, Lauer CJ, Dydak U, Hell D, Holsboer F, Boesiger P, Cuenod M. Schizophrenia: glutathione deficit in cerebrospinal fluid and prefrontal cortex in vivo. Eur J Neurosci. 2000 Oct;12(10):3721-8. doi: 10.1046/j.1460-9568.2000.00229.x. PMID 11029642
- [Background] Do KQ, Cabungcal JH, Frank A, Steullet P, Cuenod M. Redox dysregulation, neurodevelopment, and schizophrenia. Curr Opin Neurobiol. 2009 Apr;19(2):220-30. doi: 10.1016/j.conb.2009.05.001. Epub 2009 May 27. PMID 19481443
- [Background] Burgdorf JS, Christian EP, Sorensen L, Stanton PK, Leaderbrand K, Madsen TM, Khan MA, Kroes RA, Moskal JR. A translational EEG-based approach to assess modulation of long-lasting NMDAR-dependent synaptic plasticity. Psychopharmacology (Berl). 2019 Dec;236(12):3687-3693. doi: 10.1007/s00213-019-05341-w. Epub 2019 Aug 7. PMID 31392357
- See also: Study reference — https://doi.org/10.32383/appdr/89800